CLINICAL TRIAL: NCT03633084
Title: Phase 1/2 Open Label, Dose-escalation Study of the Safety and OcUlar Tolerability of a Single Intravitreal Injection of RBM-007 in Subjects witH ExudatIve Age-related Macular Degeneration (SUSHI)
Brief Title: RBM-007 in Subjects witH ExudatIve Age-related Macular Degeneration
Acronym: SUSHI
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ribomic USA Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBM-007-001
Record Dates: First submitted 2018-07-18; First posted 2018-08-16 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Intervention Model Description: This is an open label, non-controlled, sequential, dose-escalating study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- RBM-007 Injectable Solution - 0.2 mg (Experimental): No additional information.
  Interventions: Drug: RBM-007 Injectable Solution
- RBM-007 Injectable Solution - 1.0 mg (Experimental): No additional information.
  Interventions: Drug: RBM-007 Injectable Solution
- RBM-007 Injectable Solution - 2.0 mg (Experimental): No additional information.
  Interventions: Drug: RBM-007 Injectable Solution

INTERVENTIONS:
Drug: RBM-007 Injectable Solution — (No additional description)

SUMMARY:
This is an open label, non-controlled, dose-escalating study assessing the safety, tolerability, and bioactivity of a single intravitreal (i.vt.) injection of RBM-007 in approximately nine subjects with exudative age-related macular degeneration.

DETAILED DESCRIPTION:
Nine subjects in three dose cohorts (3 subjects each cohort) will receive a single i.vt. injection of RBM-007 in the study eye. Subjects will be followed through Day 56.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 55 years of age or older on the date of signing the informed consent form and able and willing to comply with all treatment and follow-up study procedures.
2. At Screening Visit, subjects must meet all the following inclusion criteria:
3. Must have had prior treatment in the study eye with any intravitreal vasoactive endothelial growth factor (VEGF) medication (at least 3 anti-VEGF) treatments within the prior 2-6 months), throughout which clinical examination and SD-OCT imaging has shown recurrent or persistent exudative activity, as shown by the presence of intraretinal or subretinal fluid, and/or subretinal exudation or hemorrhage.
4. Best corrected visual acuity of 65 to 20 Early Treatment of Diabetic Retinopathy Study (ETDRS) letters (20/50 to 20/400) in the study eye.
5. Presence of significant subretinal fluid and/or cystoid macular edema secondary to exudative age-related macular degeneration as assessed by optical coherence tomography in the study eye, with a minimum of 300 µm within the central subfield.
6. Total lesion size of ≤9 disc areas, lesion containing ≤50% hemorrhage and ≤50% subretinal fibrosis and ≤50% retinal pigment epithelial atrophy in the study eye.
7. Reasonably clear media and reasonable fixation ability in the study eye to allow for good quality tomography and fundus photography.

   At Baseline Visit (Day 0), subjects must meet all the following inclusion criteria:
8. Best Corrected Visual Acuity (BCVA) of 65 to 20 ETDRS letters (20/50 to 20/400) in the study eye.
9. Presence of significant subretinal and/or intraretinal fluid secondary to exudative age-related macular degeneration as assessed by SD-OCT in the study eye, with a minimum of 300 µm within the central subfield.
10. Total lesion size of ≤9 disc areas, containing ≤ 50% hemorrhage and ≤ 50% fibrosis and ≤ 50% retinal pigment epithelial atrophy in the study eye.

Exclusion Criteria:

Ocular exclusion criteria:

1. BCVA better than 65 ETDRS letters (20/50) in the study eye.
2. BCVA worse than 20 ETDRS letters (20/400) in study eye.
3. Fellow eye BCVA worse than 35 ETDRS letters (20/200).

   Use of any of the following treatments to the study eye:
4. Intravitreal anti-VEGF injection (ranibizumab, aflibercept or bevacizumab) in the study eye within the past 4 weeks or less prior to Baseline Visit and RBM-007 injection.
5. Intravitreal or periocular corticosteroid, within 3 months prior to Baseline Visit (Day 0) and throughout the study;
6. Fluocinolone acetonide intravitreal implant, within 12 months prior to Baseline Visit (Day 0) and throughout the study;
7. Visudyne® (verteporfin) photodynamic therapy, within 3 months prior to Baseline Visit (Day 0) and throughout the study.
8. Uncontrolled or advanced glaucoma, defined by an intraocular pressure (IOP) of >21 mmHg or cup/disc ratio > 0.8 while on medical therapy, or chronic ocular hypotony (<6 mmHg) in the study eye.
9. Evidence of ocular disease other than exudative AMD in the study eye that may confound the outcome of the study (e.g., active diabetic retinopathy, posterior uveitis, adult vitelliform dystrophy, moderate/severe myopic degeneration).
10. History of vitrectomy surgery in the study eye.
11. Anticipated need for any ocular surgery involving the study eye during the course of the study.
12. Nd:YAG laser capsulotomy within 28 days prior to Baseline Visit (Day 0) in the study eye.
13. Intraocular surgery, including lens removal or ophthalmologic laser procedure, within 90 days prior to Baseline Visit (Day 0) in the study eye.
14. Ocular or periocular infection in either eye.
15. Pupillary dilation inadequate for good quality fundus photography in the study eye.
16. Media opacity that would limit clinical visualization, fundus photography, fluorescein angiography, or SD-OCT evaluation in the study eye.
17. History of herpetic ophthalmic infection in the study eye or adnexa.
18. Presence of known toxoplasmosis or toxoplasmosis scar in either eye.
19. Presence or history of any form of ocular malignancy including choroidal melanoma in the study eye.

Ages: 55 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Ali, Ph.D., Study Director — Ribomic USA Inc
Locations (3):
- United States (3):
  - Retinal Consultants Medical Group, Sacramento, California
  - Stanford University, Stanford, California
  - Bay Area Retina Associates, Walnut Creek, California

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RBM-007 Injectable Solution - 0.2 mg | RBM-007 Injectable Solution - 1.0 mg | RBM-007 Injectable Solution - 2.0 mg
Started | 3 | 3 | 3
Completed | 3 | 3 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RBM-007 Injectable Solution - 0.2 mg | RBM-007 Injectable Solution - 1.0 mg | RBM-007 Injectable Solution - 2.0 mg | Total
Number analyzed (Participants) | 3 | 3 | 3 | 9
Age, Customized [Median (Full Range); unit: years]
  Range | 87 [71 to 88] | 80 [80 to 85] | 86 [86 to 92] | 86 [71 to 92]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 5
  Male | 2 | 2 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 3 | 9
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Ocular safety as assessed using biomicroscopy to investigate ocular tolerability [Count of Participants; unit: Participants] — Biomicroscopy is used by an ophthalmologist to assess the health of the front of the eye. The measure is the number of subjects with abnormal findings that were not present at screening. By definition, there are zero findings at baseline.
  Participants | 0 | 0 | 0 | 0
Ocular safety as assessed using ophthalmoscopy to investigate ocular tolerability [Count of Participants; unit: Participants] — Ophthalmoscopy is used by an ophthalmologist to assess the health of the back of the eye. The measure is the number of subjects with abnormal findings that were not present at screening. By definition, there are zero findings at baseline.
  Participants | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Ocular Safety as Assessed Using Biomicroscopy to Investigate Ocular Tolerability
Description: Biomicroscopy is used by an ophthalmologist to assess the health of the front of the eye. The measure is the number of subjects with abnormal findings that were not present at screening.
Time Frame: Day 56
Measure: Count of Participants; unit: Participants
Arm/Group | RBM-007 Injectable Solution - 0.2 mg | RBM-007 Injectable Solution - 1.0 mg | RBM-007 Injectable Solution - 2.0 mg
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 1

2. Primary Outcome: Ocular Safety as Assessed Using Ophthalmoscopy to Investigate Ocular Tolerability
Description: Ophthalmoscopy is used by an ophthalmologist to assess the health of the back of the eye. The measure is the number of subjects with abnormal findings that were not present at screening.
Time Frame: Day 56
Measure: Count of Participants; unit: Participants
Arm/Group | RBM-007 Injectable Solution - 0.2 mg | RBM-007 Injectable Solution - 1.0 mg | RBM-007 Injectable Solution - 2.0 mg
Number analyzed (Participants) | 3 | 3 | 3
Participants | 0 | 0 | 0

3. Secondary Outcome: Ocular Tolerability as Assessed by Number and Nature of Adverse Events
Description: Adverse events (ocular or non-ocular)
Time Frame: Day 56
Measure: Count of Participants; unit: Participants
Groups:
- RBM-007 Injectable Solution - 2 mg: No additional information.
  RBM-007 Injectable Solution: (No additional description)
Arm/Group | RBM-007 Injectable Solution - 0.2 mg | RBM-007 Injectable Solution - 1.0 mg | RBM-007 Injectable Solution - 2 mg
Number analyzed (Participants) | 3 | 3 | 3
Participants | 1 | 2 | 2

ADVERSE EVENTS:
Time Frame: 56 days
Arm/Group | RBM-007 Injectable Solution - 0.2 mg | RBM-007 Injectable Solution - 1.0 mg | RBM-007 Injectable Solution - 2.0 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 2/3 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RBM-007 Injectable Solution - 0.2 mg (N=3) | RBM-007 Injectable Solution - 1.0 mg (N=3) | RBM-007 Injectable Solution - 2.0 mg (N=3)
Subconjunctival Hemorrhage (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Mild local irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Iritis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Fall, leg injury, and sequelae (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/84/NCT03633084/Prot_SAP_001.pdf